CLINICAL TRIAL: NCT04825691
Title: ERG Protein Expression in Prostatic Acinar Adenocarcinoma and Its Correlation With Clinicopathological Features
Brief Title: ERG Protein Expression in Prostatic Adenocarcinoma and Its Clinicopathological Features
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mohammed Amin, demonstrator, Assiut University
Other Study IDs: ERG protein in cancer prostate
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases diagnosed as prostatic acinar adenocarcinoma
  Interventions: Diagnostic Test: Immunohistochemistry of prostate biopsy

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry of prostate biopsy — Sections of formalin fixed paraffin embedded tissue blocks will be stained with ERG oncoprotein. Antibody dilution, antigen retrieval methods, and incubation time will all be conducted according to the manufacturer's instructions

SUMMARY:
Evaluation the ERG expression in prostatic acinar adenocarcinoma and its association with clinicopathological features.

DETAILED DESCRIPTION:
Prostatic cancer is one of the most common malignancies in males and is the second leading cause of cancer-related deaths in males worldwide. The burden is expected to grow 1.7 million new cases and 499,000 new deaths by 2030. Although the diagnosis of prostatic carcinoma can usually be made on histological features, nowadays many immunohistochemical (IHC) markers are used to distinguish it from benign mimickers as well as in predicting prognosis and treatment. Out of these markers, Ets-related gene (ERG product) is a proto-oncogene which participates in chromosomal translocations and is frequently over expressed in prostatic carcinoma which harbors ERG-transmembrane protease, serine 2 fusion. ERG is a transcription factor belonging to the erythroblast transformation-specific (ETS) family. It is involved in many important cellular processes including differentiation, cell proliferation, angiogenesis, cell migration, hematopoiesis, and apoptosis. This proto-oncogene is expressed in the urogenital tract and hematopoietic cells. Gene fusions involving sequences of transmembrane protease serine 2 (promoter of TMPRSS2) and protein coding sequences of ERG result in over expression of ERG in prostatic tumors. This TMPRSS2-ERG fusion has been shown to occur in 50-70% cases of prostatic acinar adenocarcinoma in different studies. Genetic rearrangements were not identified in epithelial carcinomas until Tomlins et al. demonstrated ERG gene fusions in prostatic carcinoma.The presence of this fusion is now believed to be a critical event in the development of prostatic carcinoma.

TMPRSS2-ERG fusion results in constitutive expression of ERG oncoprotein resulting in enhanced proliferation and invasive potential of prostatic cancer cells. Moreover, TMPRSS2-ERG fusion gene product can be an important therapeutic target in prostatic cancer. Immunohistochemical (IHC) expression of ERG oncoprotein may serve as a surrogate biomarker of TMPRSS2-ERG fusion gene. Therefore in the present study we aimed to evaluate the ERG expression in prostatic acinar adenocarcinoma and its association with clinicopathological features.

ELIGIBILITY:
Inclusion Criteria:

* All cases diagnosed as prostatic acinar adenocarcinoma

Exclusion Criteria:

* Other types of prostatic cancer.

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All cases diagnosed as prostatic acinar adenocarcinoma.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-04 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-05-23 (Estimated)

PRIMARY OUTCOMES:
Evaluation the ERG expression in prostatic acinar adenocarcinoma | 3 days

SECONDARY OUTCOMES:
Correlation between ERG expression with clinicopathological features. | 1 week

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Clark JP, Cooper CS. ETS gene fusions in prostate cancer. Nat Rev Urol. 2009 Aug;6(8):429-39. doi: 10.1038/nrurol.2009.127. PMID 19657377
- [Background] Kumar-Sinha C, Tomlins SA, Chinnaiyan AM. Recurrent gene fusions in prostate cancer. Nat Rev Cancer. 2008 Jul;8(7):497-511. doi: 10.1038/nrc2402. Epub 2008 Jun 19. PMID 18563191
- [Background] Berg KD, Vainer B, Thomsen FB, Roder MA, Gerds TA, Toft BG, Brasso K, Iversen P. ERG protein expression in diagnostic specimens is associated with increased risk of progression during active surveillance for prostate cancer. Eur Urol. 2014 Nov;66(5):851-60. doi: 10.1016/j.eururo.2014.02.058. Epub 2014 Mar 7. PMID 24630684